CLINICAL TRIAL: NCT03350165
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Pemafibrate in Patients With Nonalcoholic Fatty Liver Disease.
Brief Title: A Study of Pemafibrate in Patients With Nonalcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kowa Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K-877-FL-01
Record Dates: First submitted 2017-11-09; First posted 2017-11-22 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — K-877 compound; (R)-2-(3-((benzoxazol-2-yl-d4 (3-(4-methoxyphenoxy-d7)propyl)amino)methyl)phenoxy) butanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): K-877 (pemafibrate) tablet twice daily.
  Interventions: Drug: K-877
- Control Group (Placebo Comparator): placebo tablet twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: K-877 — 0.2mg tablet
  Other Names: pemafibrate
  Arms: Treatment Group
Drug: Placebo — K-877 matching placebo tablet
  Arms: Control Group

SUMMARY:
A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Pemafibrate in Patients With Nonalcoholic Fatty Liver Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients show presence of hepatic fat fraction as defined by ≥ 10% on MRI-PDFF at Screening
2. Patients show presence of liver stiffness as defined by ≥ 2.5 kPa on MRE at Screening
3. Patients have an ALT above the upper limits of normal (30 IU/L for females and 40 IU/L for males) at Screening
4. Patients with NAFLD had to be age 20 years or older at written informed consent(ICF)

Exclusion Criteria:

1. Current of significant alcohol consumption (significant alcohol consumption is defined as more than 210 g/week in males and more than 140 g/week in females, on average)
2. Planned use of Contraindicated Medications from written ICF to end of treatment.
3. BMI < 22 kg/m2 at Screening
4. Uncontrolled diabetes mellitus as defined by a HbA1c(NGSP) ≥ 8.0％ at Screening
5. eGFR < 30 mL/min/1.73m2 or Dialysis patient
6. Cirrhosis
7. Biliary obstruction
8. Patients were excluded if they had evidence of other forms of liver disease shown by the following:

   * Hepatitis B or Hepatitis C
   * Autoimmune hepatitis（AIH）
   * Primary biliary cirrhosis（PBC）
   * Primary Sclerosing Cholangitis（PSC）
   * Drug-induced liver injury
   * hyperthyroidism, Wilson's disease, hemochromatosis, alpha-1-antitrypsin disease
9. Those with complicating malignant neoplasm or those judged to be at a high risk of recurrence
10. Patients with contraindications to MRI imaging
11. Patients who gave 200 mL or more of blood within 1 month before the administration of the study drug, or 400 mL or more of blood within 4 months before the administration of the study drug
12. Patients with a history of serious drug allergies (such as anaphylactic shock)
13. Pregnancy, breast feeding, planned pregnancy
14. Patients who were participating in another clinical study at the time of consent was obtained or who received study drugs other than the placebo less than 16 weeks before consent was obtained
15. Patients who have previously been administered pemafibrate
16. Patients who have been determined inappropriate by the investigator or subinvestigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Efficacy: % Change from baseline to Week 24 in hepatic fat fraction by Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI-PDFF) | Week 24
Safety: Incidence of adverse events and adverse drug reactions that occurred after the administration of the study drug | Week 24

SECONDARY OUTCOMES:
Change in noninvasive imaging biomarkers (MRI-PDFF in %, MRE in kPa, Transient elastography in kPa) | From baseline upto week 72
Change in clinical laboratory tests (AST in IU/L, ALT in IU/L, γ-GTP in IU/L) | From baseline upto week 72
Change in noninvasive biomarkers (Cytokeratin 18 in U/L, Hyaluronic acid in ng/mL, Type IV collagen 7S in ng/mL, M2BPGi in no unit) | From baseline upto week 72
Change in noninvasive biomarkers (NAFLD fibrosis score) | From baseline upto week 72
Change in noninvasive biomarkers (FIB4 index) | From baseline upto week 72
Change in noninvasive biomarkers (NAFIC score) | From baseline upto week 72
Change in noninvasive biomarkers (ELF test) | From baseline upto week 72
Percentage of patients with ≥ 30% reduction in hepatic fat fraction (MRI-PDFF) | From baseline upto week 72
Percentage of patients with ≥ 15% reduction in liver stiffness (MRE) | From baseline upto week 72

CONTACTS AND LOCATIONS:
Overall Officials: Ryohei Tanigawa, Study Director — Clinical Development Dept. Ⅰ
Locations (16):
- Japan (16):
  - Aomori Prefectural Central Hospital, Aomori, Aomori
  - Asahikawa Medical University, Asahikawa, Hokkaido
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - SeireiHamamatsu General Hospital, Hamamatsu, Shizuoka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Iwata City Hospital, Iwata, Shizuoka
  - Chutoen General Medical Center, Kakegawa, Shizuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Niigata University Medical & Dental Hospital, Niigata, Niigata
  - Ogaki Municipal Hospital, Ogaki, Gifu
  - Shiga University of Medical Science Hospital, Otsu, Shiga
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Yamagata University Hospital, Yamagata, Yamagata
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa

REFERENCES:
- [Derived] Nakajima A, Eguchi Y, Yoneda M, Imajo K, Tamaki N, Suganami H, Nojima T, Tanigawa R, Iizuka M, Iida Y, Loomba R. Randomised clinical trial: Pemafibrate, a novel selective peroxisome proliferator-activated receptor alpha modulator (SPPARMalpha), versus placebo in patients with non-alcoholic fatty liver disease. Aliment Pharmacol Ther. 2021 Nov;54(10):1263-1277. doi: 10.1111/apt.16596. Epub 2021 Sep 16. PMID 34528723
- [Derived] Fruchart JC, Hermans MP, Fruchart-Najib J, Kodama T. Selective Peroxisome Proliferator-Activated Receptor Alpha Modulators (SPPARMalpha) in the Metabolic Syndrome: Is Pemafibrate Light at the End of the Tunnel? Curr Atheroscler Rep. 2021 Jan 3;23(1):3. doi: 10.1007/s11883-020-00897-x. PMID 33392801